CLINICAL TRIAL: NCT02589054
Title: Regional Changes in Upper Limb Perfusion Following Brachial Plexus Block: A Pilot Study
Acronym: RAFFAB
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other); London Health Sciences Centre (Other); St. Joseph's Health Care London (Other)
Responsible Party: Sponsor
Other Study IDs: 106285
Record Dates: First submitted 2015-10-22; First posted 2015-10-28 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2015-10

CONDITIONS: Anesthesia, Conduction; Nerve Block; Sympathectomy; Regional Blood Flow

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients
  Interventions: Other: Monitoring

INTERVENTIONS:
Other: Monitoring

SUMMARY:
Ultrasound-guided regional anesthesia is increasingly being used in the modern surgical environment to provide specific intraoperative anesthesia and postoperative analgesia. Infiltration of local anesthesics around peripheral nerves firs blocks sympathetic, then sensory, then motor nerve function. Sympathectomy-induced vasodilation following brachial plexus block results in increased skin temperature and arterial flow within minutes.

Although it has not been shown to reliably increase diameter or cross-sectional area of distal arteries, brachial plexus block does change the pattern and quantity of blood flow to the hand. Given that the magnitude of change of flow cannot be attributed to vessel radius, the investigators suspect that the more laminar fluid dynamics are due to vascular tone.

The investigators study aims to quantify alterations in physiology and peripheral vasodilator response. The investigators anticipate that axially block will significantly improve regional blood flow.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II, III
* BMI less than or equal to 39
* Presenting for elective upper limb surgery
* Does not meet any exclusion criteria

Exclusion Criteria:

* Age over 80
* ASA physical status IV or V
* BMI greater or equal to 40
* Language barrier precluding ability to give informed consent
* History of coagulopathy
* INR < 1.4
* Platelet count < 100
* Allergy to local anesthetics
* Known peripheral vascular disease of the upper limbs
* Amputation of one or both upper limbs, not including digits
* Peripheral neurological disease
* Does not consent to participate in study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals coming for elective upper extremity surgery who would already be having a brachial plexus block for their anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in regional blood flow and perfusion characteristics in the upper arm arteries from baseline to 20 minutes after unilateral axillary block. | 30 minutes
  Physiologic parameter

SECONDARY OUTCOMES:
Changes in the caliber of the arteries of the arm between arms from baseline to 20 minutes after unilateral axillary block. | 30 minutes
  Physiologic parameter
Changes in skin temperature between hands from baseline to 20 minutes after unilateral axillary block. | 30 minutes
  Physiologic parameter
Sensory loss in radial, ulnar, and median nerve distribution between hands from baseline to 20 minutes after unilateral axillary block. | 30 minutes
  Physical examination
Motor weakness in radial, ulnar, and median nerve distributions between hands from baseline to 20 minutes after unilateral axillary block | 30 Minutes
  Physical examination